CLINICAL TRIAL: NCT06082167
Title: A Phase 2/3, Randomized, Double-Blind, Controlled Study of Zanzalintinib (XL092) in Combination With Pembrolizumab vs Pembrolizumab in First-Line Treatment of Subjects With PD-L1 Positive Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Study of Zanzalintinib (XL092) + Pembrolizumab vs Pembrolizumab in Subjects With PD-L1 Positive Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Acronym: STELLAR-305
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Exelixis (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XL092-305; KEYNOTE-G06; EU CTR: 2023-506308-24-00 (Other: European Medicines Agency); KEYNOTE-G06 (Other: Merck Sharp & Dohme LLC); MK-3475-G06 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zanzalintinib + Pembrolizumab (Experimental): Subjects with R/M HNSCC will receive zanzalintinib + pembrolizumab
  Interventions: Drug: Zanzalintinib; Biological: Pembrolizumab
- Zanzalintinib-Matched Placebo + Pembrolizumab (Placebo Comparator): Subjects with R/M HNSCC will receive zanzalintinib-matched placebo + pembrolizumab
  Interventions: Drug: Zanzalintinib-matched Placebo; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Zanzalintinib — Specified doses on specified days
  Other Names: XL092
  Arms: Zanzalintinib + Pembrolizumab
Drug: Zanzalintinib-matched Placebo — Specified doses on specified days
  Other Names: XL092-matched Placebo
  Arms: Zanzalintinib-Matched Placebo + Pembrolizumab
Biological: Pembrolizumab — Specified doses on specified days
  Other Names: KEYTRUDA®

SUMMARY:
This is a multicenter, randomized, double-blind, controlled Phase 2/3 trial of zanzalintinib in combination with pembrolizumab versus zanzalintinib-matched placebo in combination with pembrolizumab in subjects with programmed death-ligand 1 (PD-L1) positive recurrent or metastatic head and neck squamous cell carcinoma (R/M HNSCC) incurable by local therapies who have not received prior systemic therapy for recurrent or metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically-confirmed R/M HNSCC that is considered incurable by local therapy.

  * Should not have had prior systemic therapy administered in the recurrent or metastatic setting. Systemic therapy which was completed more than 6 months prior to randomization if given as part of multimodal treatment for locally advanced disease is allowed.
  * The eligible primary tumor locations are the oropharynx, oral cavity, hypopharynx, and larynx.
* PD-L1 expression level Combined Positive Score (CPS) ≥ 1.
* Participants with oropharyngeal cancer must have human papillomavirus (HPV) status from tumor tissue.
* Measurable disease according to RECIST 1.1 as determined by the Investigator.
* Tumor samples (archival or fresh tumor biopsy) are required. If archival tissue is unavailable, must provide fresh tumor tissue biopsy prior to randomization.
* Recovery to baseline or ≤ Grade 1 severity (CTCAE v5) from adverse events (AEs) related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy.
* Age 18 years (or the legal age of consent in your country, if higher than 18) or older on the day of consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Adequate organ and marrow function.

Exclusion Criteria:

* Nasopharynx, salivary gland or occult primary site (regardless of p16 status).
* Has disease that is suitable for local therapy administered with curative intent.
* Has received prior therapy with zanzalintinib, any anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (for example, cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX-40, CD137).
* Life expectancy < 3 months.
* Had progressive disease within 6 months of completion of curatively intended systemic treatment for locoregionally advanced HNSCC.
* Radiation therapy for bone metastases within 2 weeks, any other radiation therapy within 4 weeks prior to randomization.
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks prior to randomization.
* Positive hepatitis B surface antigen (HBsAg) test.
* Positive hepatitis C virus (HCV) antibody test.
* Major surgery (eg, GI surgery, removal or biopsy of brain metastasis) within 8 weeks prior to randomization. Complete wound healing from major or minor surgery must have occurred at least prior to randomization.
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 480 ms per electrocardiogram (ECG) within 28 days before randomization.
* Pregnant or lactating females.
* Administration of a live, attenuated vaccine within 30 days before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) by Blinded Independent Central Review (BICR) | Approximately 33 months after the first subject is randomized
  Defined as the time from randomization to the earlier of either radiographic progressive disease (PD) per RECIST 1.1 as determined by the BICR or death from any cause
Overall Survival (OS) | Approximately 50 months after the first subject is randomized
  Defined as the time from randomization to death due to any cause

SECONDARY OUTCOMES:
PFS per RECIST 1.1 by Investigator | Approximately 33 months after the first subject is randomized
  Defined as the time from randomization to the earlier of either radiographic PD per RECIST 1.1 as determined by the Investigator or death from any cause
Objective Response Rate (ORR) per RECIST 1.1 by the BICR and Investigator | Approximately 33 months after the first subject is randomized
  Defined as the proportion of subjects with the best overall response of complete response (CR) or partial response (PR) per RECIST 1.1 as determined by the BICR and Investigator
Duration of Response (DOR) Per RECIST 1.1 by BICR and Investigator | Approximately 33 months after the first subject is randomized
  Defined as the time from the first documentation of objective response (subsequently confirmed at a visit ≥ 28 days later) to disease progression or death due to any cause

CONTACTS AND LOCATIONS:
Locations (168):
- United States (15):
  - Exelixis Clinical Site #2, Fullerton, California
  - Exelixis Clinical Site #1, Orange City, Florida
  - Exelixis Clinical Site #163, Tampa, Florida
  - Exelixis Clinical Site #123, Athens, Georgia
  - Exelixis Clinical Site #82, Atlanta, Georgia
  - Exelixis Clinical Site #19, Chicago, Illinois
  - Exelixis Clinical Site #62, Des Moines, Iowa
  - Exelixis Clinical Site #100, Iowa City, Iowa
  - Exelixis Clinical Site #4, St Louis, Missouri
  - Exelixis Clinical Site #148, Lebanon, New Hampshire
  - Exelixis Clinical Site #158, Camden, New Jersey
  - Exelixis Clinical Site #3, Shirley, New York
  - Exelixis Clinical Site #95, Durham, North Carolina
  - Exelixis Clinical Site #117, Wilson, North Carolina
  - Exelixis Clinical Site #43, Roanoke, Virginia
- Argentina (8):
  - Exelixis Clinical Site #73, Rosario, Santa Fe Province
  - Exelixis Clinical Site #91, Buenos Aires
  - Exelixis Clinical Site # 47, Ciudad Autonoma de Buenos Aire
  - Exelixis Clinical Site #53, Ciudad Autonoma de Buenos Aire
  - Exelixis Clinical Site #93, Córdoba
  - Exelixis Clinical Site #64, Córdoba
  - Exelixis Clinical Site #157, Pergamino
  - Exelixis Clinical Site #92, Santa Fe
- Australia (5):
  - Exelixis Clinical Site #57, Port Macquarie, New South Wales
  - Exelixis Clinical Site # 46, Adelaide
  - Exelixis Clinical Site #154, Bedford Park
  - Exelixis Clinical Site #137, Camperdown
  - Exelixis Clinical Site #39, Murdoch
- Austria (3):
  - Exelixis Clinical Site #156, Linz
  - Exelixis Clinical Site #42, Salzburg
  - Exelixis Clinical Site #166, Vienna
- Belgium (4):
  - Exelixis Clinical Site #22, Brussels
  - Exelixis Clinical Site #106, Charleroi
  - Exelixis Clinical Site #14, Libramont
  - Exelixis Clinical Site #37, Sint-Niklaas
- Brazil (16):
  - Exelixis Clinical Site #68, Passo Fundo, Rio Grande do Sul
  - Exelixis Clinical Site #90, Porto Alegre, Rio Grande do Sul
  - Exelixis Clinical Site #110, Jaú, São Paulo
  - Exelixis Clinical Site #65, Santo André, São Paulo
  - Exelixis Clinical Site #83, São José do Rio Preto, São Paulo
  - Exelixis Clinical Site #116, Barretos
  - Exelixis Clinical Site #75, Curitiba
  - Exelixis Clinical Site #101, Curitiba
  - Exelixis Clinical Site #97, Porto Alegre
  - Exelixis Clinical Site #102, Recife
  - Exelixis Clinical Site #87, Rio de Janeiro
  - Exelixis Clinical Site #76, São Paulo
  - Exelixis Clinical Site #77, São Paulo
  - Exelixis Clinical Site #67, São Paulo
  - Exelixis Clinical Site #98, São Paulo
  - Exelixis Clinical Site #88, São Paulo
- Bulgaria (5):
  - Exelixis Clinical Site #25, Plovdiv
  - Exelixis Clinical Site #94, Rousse
  - Exelixis Clinical Site #15, Sofia
  - Exelixis Clinical Site #11, Sofia
  - Exelixis Clinical Site #54, Sofia
- Chile (7):
  - Exelixis Clinical Site #33, Santiago
  - Exelixis Clinical Site #52, Santiago
  - Exelixis Clinical Site #38, Santiago
  - Exelixis Clinical Site #109, Santiago
  - Exelixis Clinical Site #50, Talca
  - Exelixis Clinical Site #51, Valdivia
  - Exelixis Clinical Site #40, Viña del Mar
- Colombia (5):
  - Exelixis Clinical Site #96, Barranquilla
  - Exelixis Clinical Site #152, Bogotá
  - Exelixis Clinical Site #103, Floridablanca
  - Exelixis Clinical Site #146, Pasto
  - Exelixis Clinical Site #149, Pereira
- Czechia (6):
  - Exelixis Clinical Site #49, Nový Jičín
  - Exelixis Clinical Site #58, Olomouc
  - Exelixis Clinical Site #151, Prague
  - Exelixis Clinical Site #34, Prague
  - Exelixis Clinical Site #48, Prague
  - Exelixis Clinical Site #36, Prague
- France (13):
  - Exelixis Clinical Site #28, Marseille, Bouches-du-Rhône
  - Exelixis Clinical Site #16, Bordeaux, Gironde
  - Exelixis Clinical Site #44, Rennes, Ille Et Vilaine
  - Exelixis Clinical Site #108, Saint Priest En Jarez, Pays de la Loire Region
  - Exelixis Clinical Site #70, Lyon, Rhone
  - Exelixis Clinical Site #107, Le Mans, Sarthe
  - Exelixis Clinical Site #66, Villejuif, Val De Marne
  - Exelixis Clinical Site #144, Dijon
  - Exelixis Clinical Site #141, Grenoble
  - Exelixis Clinical Site #140, Lille
  - Exelixis Clinical Site #26, Paris
  - Exelixis Clinical Site #112, Pierre-Bénite
  - Exelixis Clinical Site #105, Poitiers
- Exelixis Clinical Site #167, Giessen, Germany
- Greece (6):
  - Exelixis Clinical Site #155, Athens
  - Exelixis Clinical Site #129, Athens
  - Exelixis Clinical Site #159, Larissa
  - Exelixis Clinical Site #120, Thessaloniki
  - Exelixis Clinical Site #150, Thessaloniki
  - Exelixis Clinical Site #128, Thessaloniki
- Hungary (4):
  - Exelixis Clinical Site #125, Budapest
  - Exelixis Clinical Site #99, Kecskemét
  - Exelixis Clinical Site #131, Salgótarján
  - Exelixis Clinical Site #147, Szekszárd
- Israel (5):
  - Exelixis Clinical Site #132, Haifa
  - Exelixis Clinical Site #85, Haifa
  - Exelixis Clinical Site #74, Jerusalem
  - Exelixis Clinical Site #122, Ramat Gan
  - Exelixis Clinical Site #86, Tel Aviv
- Italy (9):
  - Exelixis Clinical Site #21, Candiolo, Torino
  - Exelixis Clinical Site #35, Brescia
  - Exelixis Clinical Site #45, Catania
  - Exelixis Clinical Site #81, Milan
  - Exelixis Clinical Site #55, Milan
  - Exelixis Clinical Site #18, Napoli
  - Exelixis Clinical Site #78, Rome
  - Exelixis Clinical Site #124, Rozzano
  - Exelixis Clinical Site #10, Verona
- Malaysia (3):
  - Exelixis Clinical Site #61, Putrajaya, Kuala Lumpur
  - Exelixis Clinical Site #60, Kuala Lumpur
  - Exelixis Clinical Site #72, Kuala Lumpur
- Mexico (3):
  - Exelixis Clinical Site #114, Guadalajara, Jalisco
  - Exelixis Clinical Site #119, San Juan del Río, Querétaro
  - Exelixis Clinical Site #168, Guadalajara
- Poland (3):
  - Exelixis Clinical Site #89, Piotrków, Trybunalski
  - Exelixis Clinical Site #139, Gliwice
  - Exelixis Clinical Site #162, Torun
- Romania (6):
  - Exelixis Clinical Site #160, Bucharest
  - Exelixis Clinical Site #24, Cluj-Napoca
  - Exelixis Clinical Site #20, Craiova
  - Exelixis Clinical Site #104, Floreşti
  - Exelixis Clinical Site #127, Ploieşti
  - Exelixis Clinical Site #143, Timișoara
- Slovakia (3):
  - Exelixis Clinical Site #23, Košice
  - Exelixis Clinical Site #27, Trnava
  - Exelixis Clinical Site #121, Žilina
- South Korea (12):
  - Exelixis Clinical Site #7, Busan, Gangwon-do
  - Exelixis Clinical Site #30, Suwon, Gyeonggi-do
  - Exelixis Clinical Site #17, Suwon, Gyeonggi-do
  - Exelixis Clinical Site #9, Yangsan, Gyeongsangnam-do
  - Exelixis Clinical Site #69, Jeonju, Jeollabuk-do
  - Exelixis Clinical Site #8, Jeonju, Jeollabuk-do
  - Exelixis Clinical Site #13, Busan
  - Exelixis Clinical Site #5, Seoul
  - Exelixis Clinical Site #63, Seoul
  - Exelixis Clinical Site #12, Seoul
  - Exelixis Clinical Site #6, Seoul
  - Exelixis Clinical Site #29, Seoul
- Spain (12):
  - Exelixis Clinical Site #130, A Coruña
  - Exelixis Clinical Site #115, Barcelona
  - Exelixis Clinical Site #113, Girona
  - Exelixis Clinical Site #134, Madrid
  - Exelixis Clinical Site #111, Madrid
  - Exelixis Clinical Site #32, Madrid
  - Exelixis Clinical Site #59, Madrid
  - Exelixis Clinical Site #31, Madrid
  - Exelixis Clinical Site #136, Pamplona
  - Exelixis Clinical Site #126, Seville
  - Exelixis Clinical Site #153, Valencia
  - Exelixis Clinical Site #41, Zaragoza
- Taiwan (5):
  - Exelixis Clinical Site #145, Kaohsiung City
  - Exelixis Clinical Site #164, Taichung
  - Exelixis Clinical Site #118, Taipei
  - Exelixis Clinical Site #142, Taipei
  - Exelixis Clinical Site #165, Taoyuan District
- Thailand (4):
  - Exelixis Clinical Site #71, Bangkoknoi, Bangkok
  - Exelixis Clinical Site #79, Hat Yai, Changwat Songkhla
  - Exelixis Clinical Site #56, Chiang Mai, Chiang Mai
  - Exelixis Clinical Site #80, Bangkok
- United Kingdom (5):
  - Exelixis Clinical Site #135, London, England
  - Exelixis Clinical Site #84, Romford, Essex
  - Exelixis Clinical Site #138, Manchester
  - Exelixis Clinical Site #133, Sutton
  - Exelixis Clinical Site #161, Torquay

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saba NF, Harrington K, Licitra L, Machiels JP, He C, Jew T, Andrianov V, Haddad R. STELLAR-305: phase II/III study of zanzalintinib plus pembrolizumab versus pembrolizumab alone in patients with HNSCC. Future Oncol. 2025 May;21(11):1349-1356. doi: 10.1080/14796694.2025.2485015. Epub 2025 Apr 18. PMID 40248950